CLINICAL TRIAL: NCT06525649
Title: A Double Blind, Randomized, Cross-over Study Examining the Suppression of the Photoparoxysmal EEG Response With NPT 2042
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeuroPro Therapeutics, Inc. (Industry)
Collaborators: The Epilepsy Study Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: NPT 2042 CL-102
Record Dates: First submitted 2024-07-15; First posted 2024-07-29 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Photosensitive Epilepsy; Epilepsy
MeSH Terms: conditions — Epilepsy, Reflex; Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The subject, investigator, staff, and EEG adjudicator will be blinded to the treatment assignment. All sponsor personnel will be unblinded except the sponsor's study monitor who will remain blinded.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Matching placebo for active comparator.
  Interventions: Drug: NPT 2042
- NPT 2042 160mg (Active Comparator): NPT 2042
  Interventions: Drug: NPT 2042
- NPT 2042 240mg (Active Comparator): NPT 2042
  Interventions: Drug: NPT 2042

INTERVENTIONS:
Drug: NPT 2042 — NPT 2042 is a new drug being developed as an anti-seizure treatment.

SUMMARY:
A double-blind, placebo-controlled, crossover trial to investigate the PPR of approximately 5 subjects with a known stable PPR on EEG, using 2 doses of NPT 2042 compared to placebo.

DETAILED DESCRIPTION:
This study will compare the effect of 2 doses of NPT 2042 on the photoparoxysmal- electroencephalogram (EEG) response (PPR), compared to placebo. Subjects will be screened to ensure they have a stable PPR. Subjects will then return for 3 treatment visits, each lasting 1 day, with minimum 14-day washout period between visits. Subjects will be randomized to a treatment sequence in order to receive NPT 2042 (160 mg or 240 mg) or matching placebo on each treatment day. The PPR will be measured at predose (-0.5 hours) and 0.5, 1, 2, 3, 4, and 6 hours postdose. The PPR of the active treatments will be compared to the placebo response.

ELIGIBILITY:
Inclusion Criteria:

1. Subject or legal authorized representative/guardian must be able to provide written informed consent signed prior to any study-specific procedures being conducted.
2. Individuals aged 18-75 years at the time of consent.
3. Subject has a diagnosis and history of a PPR with or without a diagnosis of epilepsy.
4. Subjects receiving zero to three concomitant antiseizure medications (ASMs).

   * Benzodiazepines: the chronic use of a benzodiazepine for any indication will be allowed and will be counted as an ASM.
   * Vagus nerve stimulator (VNS)/responsive neurostimulation (RNS): VNS/RNS will not be counted toward the number of concomitant ASMs. Subjects with surgically implanted VNS/RNS will be allowed to enter the study if all the following conditions are met:

     * The device has been in place for 1 year or more prior to the screening visit.
     * The settings have remained constant for 3 months or more prior to the screening visit and remain constant throughout the study.
     * The battery is expected to last for the duration of the study.
5. At least 3 of the EEGs performed during the screening visit must have an intermittent photic stimulation (IPS)-induced SPR of ≥3 points on a frequency assessment scale in the same eye condition, with documented confirmation by the Epilepsy Study Consortium, Inc. (ESCI).
6. Subject is in otherwise good health (with the exception of epilepsy), as determined by the investigator and documented in the medical history.
7. Subject has a body mass index (BMI) between 18 and 40 kg/m2.
8. Subject agrees to refrain from strenuous exercise which is not within the subject's normal daily routine the day before screening, as determined by the investigator.
9. Female subjects of childbearing potential and all men: agree to use of highly effective methods of contraception during the study and for 28 days after last dose of study drug.
10. Subject is able to communicate with the investigator and to understand and comply with all study requirements.

Exclusion Criteria:

1. Subject has a history of non-epileptic seizures (e.g., metabolic, structural, or pseudoseizures).
2. Females who are pregnant or lactating.
3. Subject has a clinically significant laboratory abnormality that, in the opinion of the investigator, will exclude the subject from the study.
4. Subject has an active central nervous system (CNS) infection, demyelinating disease, degenerative neurological disease, or any CNS disease deemed to be progressive during the course of the study that may confound the interpretation of the study results.
5. Subject has any clinically significant psychiatric illness, psychological, or behavioral problems which, in the opinion of the investigator, would interfere with the subject's ability to participate in the study.
6. Subject has clinically significant active liver disease (i.e., liver function tests greater than 3 times the upper limit of normal aspartate aminotransferase (AST), or alanine aminotransferase (ALT), porphyria, or has a family history of severe hepatic dysfunction.
7. Subject has a history of alcoholism, drug abuse, or drug addiction within the past 12 months.
8. Subjects who have participated in any other trials involving an investigational product or device within 30 days or five half-lives (whichever is longer) of Screening.
9. Subject is currently using of any prohibited medication, food or supplement
10. Inability of the investigator to reliably distinguish between spontaneous and provoked spike-wave burst discharges.
11. Subject uses a benzodiazepine as rescue medication within 24 hours of screening. If, in the judgment of the investigator, the subject meets all of the inclusion and none of the other exclusion criteria, rescreening may be done after appropriate wash-out period. If no other rescue medications have been used within the past month, the subject may be eligible for rescreening.
12. Subject has more than one use of rescue medications in the past 30 days.
13. Subject has a history of suicidal thoughts or behaviors in the past 6 months or more than one lifetime suicide attempt.
14. Subject is unable to complete ingestion of 12 placebo SGCs with a minimum of 8 ounces of water at screening.
15. Subject has a clinically significant medical condition that would interfere with the subject's ability to participate in the study (e.g. active cancer, cardiac disease, renal insufficiency, or active infectious processes).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-08-21 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Evaluate the change in the adjudicated SPR (standard photosensitivity range) | Through study completion, an average of 4 months
  Evaluate the change in the adjudicated SPR (standard photosensitivity range) in subjects receiving each different dose strengths of NPT 2042 compared to placebo in the most sensitive eye condition. The most sensitive eye condition will be determined at the screening visit.

SECONDARY OUTCOMES:
Change in adjudicated SPR | Through study completion, an average of 4 months
  Evaluate the change in adjudicated SPR in subjects receiving each dose strength of NPT 2042 compared to placebo in all eye conditions.
Explore the time of PPR effect to the NPT 2042 and metabolite plasma concentration-time profiles in the most sensitive eye condition. | Through study completion, an average of 4 months
  Explore the time of PPR effect to the NPT 2042 and metabolite plasma concentration-time profiles in the most sensitive eye condition.
Explore the onset of PPR effect to the NPT 2042 and metabolite plasma concentration-time profiles in all eye conditions. | Through study completion, an average of 4 months
  Explore the onset of PPR effect to the NPT 2042 and metabolite plasma concentration-time profiles in all eye conditions.
Explore the duration of PPR effect to the NPT 2042 and metabolite plasma concentration-time profiles in all eye conditions. | Through study completion, an average of 4 months
  Explore the duration of PPR effect to the NPT 2042 and metabolite plasma concentration-time profiles in all eye conditions.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Trials, Inc. (CTI), Little Rock, Arkansas
  - Idaho Comprehensive Epilepsy Center, Boise, Idaho